CLINICAL TRIAL: NCT05839418
Title: Sustained Effort Network for Treatment of Status Epilepticus/European Academy of Neurology Registry on Refractory Status Epilepticus (SENSE-II/AROUSE)
Acronym: SENSEII/AROUSE
Status: Recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2020/483/B4062020000170
Record Dates: First submitted 2023-03-23; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-03

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SENSE-II/AROUSE is a prospective, multicenter registry for patients treated for SE. The primary objective is to document patients and SE characteristics, treatment modalities, EEG features, and outcome of consecutive adults admitted fir SE treatment in each of the participating centers and to identify predictors of outcome and refractoriness.

DETAILED DESCRIPTION:
SENSE-II/AROUSE is a prospective, multicenter, non-randomized, observational registry study of consecutive cases of SE. We aimed to include university hospitals as well as non-university hospitals to enhance generalizability of the findings.

Currently, 13 high-volume medical centers in Belgium, Austria, Germany, United Kingdom, Switzerland, No common management protocol will be imposed on the participating centers. However, most institutions have established a local protocol that is closely related to the most recent guidelines for the management of SE published by the American Epilepsy Society (AES) in 2016.

We will exclude patients with anoxic status epilepticus after cardiac arrest and patients younger than 18 years.

Clinical and EEG Data will be collected prospectively from the admission of the patient to the discharge. Data collection will be performed using Research Electronic Data Capture (REDCap) electronic data capture tools hosted at Erasme Hospital in Brussels, Belgium.

To reach sufficient statistical power for multivariate analysis, a cohort size of 3000 patients is targeted.

The main objective of the study is to document patient characteristics, treatment modalities, EEG features and outcome of adults treated for SE and identify predictors of outcome. The data collected in this study could also identify gaps and opportunities for the management of this medical emergency. Lacking adequate prospective controlled trials, this will help both decision-making in clinical practice and designing future clinical trials.

Moreover, EEG data will help for a better electroencephalographic definition of SE, possible SE, and some boundary conditions, such as ictal-interictal continuum.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above
* Patients admitted for management of Status Epilepticus as their primary diagnosis
* Patients admitted for another primary diagnosis but identified with Status Epilepticus during their acute hospital stay

Exclusion Criteria:

- Patients with post-cardiac arrest SE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of and above 18 years admitted for Status Epilepticus management or who develop Status Epilepticus during their hospital stay
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | On the date of discharge from hospital or date of death from any cause, assessed up to 24 months
  Functional outcome will be assessed by the modified Rankin scale (mRS). mRS is as scale from 0 to 6 : 0 being a patient without symptoms (better outcome) and 6 being a deceased patient (worse outcome).
Refractoriness | From date of study inclusion until the date of discharge from hospital or date of death from any cause, assessed up to 24 months
  Refractory Status Epilepticus is defined as Status Epilepticus persisting despite administration of at least two appropriately selected and dosed parenteral medications including a benzodiazepine.

SECONDARY OUTCOMES:
Modified Rankin Scale | At 30 days after the date of inclusion or SE onset (if still hospitalized)
  Functional outcome will be assessed by the modified Rankin scale (mRS). mRS is as scale from 0 to 6 : 0 being a patient without symptoms (better outcome) and 6 being a deceased patient (worse outcome).
Modified Rankin Scale | At 3 months after the date of discharge from hospital
  Functional outcome will be assessed by the modified Rankin scale (mRS). mRS is as scale from 0 to 6 : 0 being a patient without symptoms (better outcome) and 6 being a deceased patient (worse outcome).
Super-refractoriness | From date of study inclusion until the date of discharge from hospital or date of death from any cause, assessed up to 24 months
  Super-refractory status epilepticus is defined as Status Epilepticus persisting or recurring after 24 hours or more of treatment with continuous intravenous anesthetic drugs or when therapy is tapered after 24 hours of use.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Gaspard, MD, PhD, Principal Investigator — Erasme UH
Locations (11):
- Austria (2):
  - Kepler University Linz, Linz
  - Christian Doppler Klinik of Paracelsus Medical University, Salzburg
- HUB Erasme, Brussels, Belgium
- Odense University Hospital & Svenborg Hospital, Odense, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- Germany (2):
  - Goethe-Universität Frankfurt am Main, Frankfurt
  - Epilepsy Center Münster-Osnabrück, Klinikum Osnabrück, Osnabrück
- Oslo University Hospital, Oslo, Norway
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital of Geneva, Geneva
- Birmingham University Hospitals NHS Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared with other researchers. not public upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be deidentified and collected through RedCap by each local investigator.
  IPD will be accessible and shared only with the researchers involved in this registry.
  These de-identified data will be available for the duration of the registry and on reasonable request to Nicolas Gaspard after publication of the results.
Access Criteria: IPD will be accessible only by the researchers involved in the building of this registry.

REFERENCES:
- [Derived] Damien C, Leitinger M, Kellinghaus C, Strzelczyk A, De Stefano P, Beier CP, Sutter R, Kamppi L, Strbian D, Tauboll E, Rosenow F, Helbok R, Ruegg S, Damian M, Trinka E, Gaspard N. Sustained effort network for treatment of status epilepticus/European academy of neurology registry on adult refractory status epilepticus (SENSE-II/AROUSE). BMC Neurol. 2024 Jan 4;24(1):19. doi: 10.1186/s12883-023-03505-y. PMID 38178048